CLINICAL TRIAL: NCT00755443
Title: A Randomized Comparison of Sirolimus-Eluting Stent Versus Standard Stent for Percutaneous Coronary Revascularization in Diabetic Patients
Brief Title: Sirolimus-Eluting Stent Versus Standard Stent in Diabetic
Acronym: DIABETES
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital San Carlos, Madrid (Other)
Collaborators: Hospital Clínico Universitario de Valladolid (Other); Hospital Universitari de Bellvitge (Other); Hospital de Meixoeiro (Other Government)
Responsible Party: Manel Sabate, Hospital Clinico San Carlos
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DIABETES I TRIAL
Record Dates: First submitted 2008-09-18; First posted 2008-09-19 (Estimated); Last update posted 2008-09-19 (Estimated); Status verified 2008-09

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Drug-Eluting Stents

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Experimental)
  Interventions: Device: Drug eluting stent
- 1 (Placebo Comparator): Bare metal stent
  Interventions: Device: Bare metal stent

INTERVENTIONS:
Device: Drug eluting stent — Drug eluting stent implantation
  Arms: 2
Device: Bare metal stent
  Arms: 1

SUMMARY:
The purpose of this study was to determine whether Sirolimus stent implantation is effective in reducing neointimal hyperplasia as compared to Bare metal stent in diabetic patients with de novo coronary artery stenosis.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic either non-insulin or insulin-dependent (according to World Health Organization Report) on pharmacologic treatment (insulin or hypoglycaemic agents) for at least 1 month, and presented de novo coronary stenoses in 1,2 or 3 native vessels with symptoms or objective evidence of ischemia. Stenoses had to be amenable for stent implantation, with vessel size smaller than 4.0 mm (as assessed visually on angiography)

Exclusion Criteria:

* Impaired glucose tolerance without pharmacologic treatment, gestational diabetes or transient hyperglycaemia
* Stenoses located in saphenous bypass, arterial bypass grafting, unprotected left main or involving important side branches (> 2 mm) that should be treated during the procedure
* Left ventricle ejection fraction < 25%
* Prior treatment with intracoronary brachytherapy or other drug eluting stent at target site
* Restenotic lesions; known allergies to aspirin, ticlopidine and clopidogrel acute coronary syndromes with persistent ST elevation < 72 hours and/or CPK twice the upper normal limit
* Non-ST elevation acute coronary syndromes with CPK twice the upper normal limit
* Severe hepatic or renal disease (creatinin clearance < 30 ml/min or hepatic enzymes twice the upper normal limit); and life expectancy < 1 year

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2003-02; Primary Completion 2004-09 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of this study was in-segment late lumen loss as assessed by quantitative coronary angiography | 270-day follow-up

SECONDARY OUTCOMES:
Other angiographic parameters of restenosis such as binary restenosis, and minimal luminal diameter; major adverse cardiac events including cardiac death, myocardial infarction, target lesion (in-segment zone) revascularization stent thrombosis | 1, 9, 12 and 24-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Manel Sabate, Md, PhD, Principal Investigator — Hospital Clinico San Carlos
Locations (1):
- Hospital Clinico San carlos, Madrid, Madrid, Spain

REFERENCES:
- [Result] Sabate M, Jimenez-Quevedo P, Angiolillo DJ, Gomez-Hospital JA, Alfonso F, Hernandez-Antolin R, Goicolea J, Banuelos C, Escaned J, Moreno R, Fernandez C, Fernandez-Aviles F, Macaya C; DIABETES Investigators. Randomized comparison of sirolimus-eluting stent versus standard stent for percutaneous coronary revascularization in diabetic patients: the diabetes and sirolimus-eluting stent (DIABETES) trial. Circulation. 2005 Oct 4;112(14):2175-83. doi: 10.1161/CIRCULATIONAHA.105.562421. PMID 16203930